CLINICAL TRIAL: NCT00209534
Title: A Phase 2, Two Part Study of AQUAVAN® Injection in the Presence of Pre-Medication in Patients Undergoing Elective Colonoscopy
Brief Title: A Study of AQUAVAN® Injection in the Presence of Pre-Medication in Patients Undergoing Elective Colonoscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Omnicare Clinical Research (Industry); Bio Analytical Research Corporation (Industry); MDS Pharma Services (Industry); The Coghlan Group (Plasma Sample Supplies) (Unknown); HHI Clinical Research (Biostatistics) (Unknown)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 3000-0207
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2009-12-04 (Estimated); Status verified 2009-12

CONDITIONS: Colonoscopy; Colon Polyps
MeSH Terms: conditions — Colonic Polyps | interventions — fospropofol

INTERVENTIONS:
Drug: fospropofol disodium

SUMMARY:
This study was designed to assess the safety and efficacy of AQUAVAN® Injection in providing adequate sedation in patients undergoing colonoscopy. Prior to the procedure, patients received fentanyl citrate for pain management followed five minutes later by AQUAVAN® Injection for sedation. Throughout the procedure, study personnel assessed the patient's vital signs and depth of sedation. After the procedure, the patient, physician, and an evaluator were asked to complete satisfaction surveys.

DETAILED DESCRIPTION:
Randomized, open label, multi-center, adaptive dose ranging study, in which several dose levels of AQUAVAN® Injection and fentanyl citrate injection will be investigated to produce a desired sedation level in patients undergoing elective colonoscopy. A desired sedative dose/dose range and dosing paradigm will be identified based on pre-set criteria using the Modified Observer's Assessment of Alertness/Sedation (OAA/S). The desired sedative dose/dose range and dosing paradigm of AQUAVAN® Injection is defined as one that consistently provides mild to moderate sedation (Modified OAA/S between 2 and 4 inclusive) in a majority of patients who are pre-medicated with fentanyl citrate injection.

ELIGIBILITY:
Inclusion Criteria:

1. Patients provided written informed consent after receiving a full explanation of the extent and nature of the study.
2. Patients were >=18 years of age to ≤60 years (a subset of up to 50 patients >60 years and <85 years of age was allowed).
3. Patients, if female, were surgically sterile, postmenopausal or non-pregnant using an acceptable method of birth control for at least 1 month prior to dosing, with a negative urine pregnancy test result at screening and predose.
4. Body mass index (BMI) between 20 and 28.
5. Body weight between 50 kg and 100 kg.
6. Patients had an ASA Physical Classification System status of I or II;
7. Patients required an elective colonoscopy procedure that was anticipated to be performed in <60 minutes (i.e., procedure was predicted to be uncomplicated); desired sedation for the colonoscopy procedure; and were determined by the Investigator to be physically capable of maintaining an adequate airway during mild-to-moderate sedation.

Exclusion Criteria:

1. Patients ingested benzodiazepines or barbiturates within 14 days of study start, with the exception of phenobarbital, which required a 21-day washout.
2. Patients ingested opioids within 72 hours of study start.
3. Patients had current symptoms of upper respiratory infection.
4. Patients had a history of allergic reaction or hypersensitivity to any anesthetic agent, narcotic, or benzodiazepine.
5. Patients had current signs of significant hiatal hernia, esophageal reflux, or heartburn which, in the opinion of the Investigator, could interfere with maintenance of an adequate airway.
6. Patients had a history of alcohol or drug abuse within the past 12 months;
7. Patients ingested alcohol or caffeine within 12 hours prior to admission into the study.
8. Patients participated in an investigational drug study within 1 month prior to study start.
9. Patients were unwilling to adhere to preprocedural and postprocedural instructions.
10. Patients donated >300 mL of blood within 1 month prior to study start; or
11. Patients were exposed to AQUAVAN in a previous clinical trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2003-01; Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
The primary efficacy objective was to determine the desired sedative dose/dose range and dosing paradigm of AQUAVAN, defined as one that consistently provided mild-to-moderate sedation (Modified OAA/S >=2 and <=4) in a majority of patients.

SECONDARY OUTCOMES:
Efficacy variables included: time to sedation, time to Fully Alert, time to Fully Recovered, time to Ready for Discharge, Modified OAA/S scores over time, number of doses and amount of AQUAVAN, and Patient and Physician Satisfaction Surveys.

CONTACTS AND LOCATIONS:
Overall Officials: James Jones, MD,PharmD, Study Director — Eisai Inc.